CLINICAL TRIAL: NCT02714725
Title: Effect Of Dexmedetomidine Infusion On Sublingual Microcirculation In Patients Undergoing On Pump Coronary Artery Bypass Graft Surgery
Brief Title: Effect Of Dexmedetomidine On Sublingual Microcirculation In Patients Undergoing On Pump CABG Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan mohamed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-54-2015
Record Dates: First submitted 2016-03-13; First posted 2016-03-21 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Sublingual Microcirculation
Keywords: Dexmedetomidine; Microcirculation; On Pump; CABG
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Group C) (Placebo Comparator): During bypass, patients in this group will receive propofol infusion 50 - 70 mcg/kg/min plus normal saline infusion
  Interventions: Drug: Placebo for Dexmedetomidine normal saline infusion; Drug: Propofol infusion
- Group Dexmedetomidine (Group DEX) (Active Comparator): During bypass, patients in this group will receive propofol infusion 50 - 70 mcg/kg/min plus dexmedetomidine infusion 0.5 mcg/kg/hr
  Interventions: Drug: Dexmedetomidine; Drug: Propofol infusion

INTERVENTIONS:
Drug: Dexmedetomidine — During bypass, patients will receive dexmedetomidine infusion 0.5 mcg/kg/hr
  Other Names: Precedex
  Arms: Group Dexmedetomidine (Group DEX)
Drug: Placebo for Dexmedetomidine normal saline infusion — During bypass, patients will receive normal saline infusion
  Other Names: Normal saline infusion
  Arms: Control group (Group C)
Drug: Propofol infusion — During bypass, patients will receive propofol infusion 50 - 70 mcg/kg/min
  Other Names: Diprivan

SUMMARY:
This study is designed to explore the possible effects of dexmedetomidine infusion on sublingual microcirculation in patients undergoing on-pump coronary artery bypass graft surgery

DETAILED DESCRIPTION:
All patients will be premedicated the night before surgery with bromazepam 3 mg PO, and 0.1 mg/Kg morphine sulphate IM one hour preoperatively. Upon arrival to the pre-induction room, the patient will receive supplementary oxygen via a nasal cannula, and will be monitored with ECG, Non invasive blood pressure and pulse oximeter. Under local infiltration anesthesia (lidocaine 2%) a peripheral venous cannula (14 or 16 G) and a 20 G arterial cannula will be inserted. Induction of anesthesia will be accomplished with fentanyl (7-10 μg/Kg), propofol 0.5 - 1.0 mg/Kg and pancuronium (0.08 - 0.12 mg/Kg). After intubation a triple lumen central venous catheter will be inserted in a central vein. The temperature probe will be inserted in the nasopharynx; the TEE probe will be also inserted after decompression of the stomach with a nasogastric tube.

All patients will be mechanically ventilated with a tidal volume of 6-8 mL/kg and a respiratory rate of 12 - 14 to achieve end-tidal CO2 30 - 35 mmHg . A PEEP of 5 cm H2O is also added. FiO2 will be adjusted to achieve a PaO2 between 200 and 300 mmHg. Isoflurane will be adjusted to 1 - 1.5 expired MAC , as well as fentanyl increments of 2 μg/Kg will be used to control adequate level of anesthesia and to maintain hemodynamic stability. Incremental doses of pancuronium will be administered as needed.

Before starting CPB anticoagulation with 400IU/kg heparin iv will be administered and activated clotting time (ACT) will be used to check proper anticoagulation throughout CPB aiming at ACT >400s.

Cardiopulmonary bypass flow rate of 2.2 - 2.4 l/min/m2 is maintained aiming to keep MAP of 50-80 mmHg together with the use of vasopressors and vasodilators when needed. After Initiation of CPB mild hypothermia (34-35℃) will be performed . During weaning from CPB, volume and pharmacological therapy with inotropes and vasodilators will be used as needed to maintain hemodynamic stability. All blood on the CPB machine will be re-infused into the patient and protamine will be administered in a dose of 4 mg/kg to return ACT to baseline values.

Using a computer-generated random sequence of numbers, patients will be allocated to one of the following two study groups:

- Control group (Group C): During bypass, patients in this group will receive propofol infusion 50 - 70 mcg/kg/min plus normal saline infusion

- Group Dexmedetomidine (Group DEX): During bypass, patients in this group will receive propofol infusion 50 - 70 mcg/kg/min plus dexmedetomidine infusion 0.5 mcg/kg/hr Patients and investigators performing the study and assessing its outcomes will all be blinded to the study group allocation. The study drugs will be prepared by a separate investigator not involved in either study performance or analysis.

Data collection Microcirculation will be studied with side-stream dark field (SDF) imaging (Microscan; MicroVision Medical, Amsterdam, Netherlands) at three times; Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass (T2) Side stream dark field imaging is equipped with sterile caps to avoid contamination. Briefly, after gentle cleansing by isotonic-saline-drenched gauze, avoiding pressure artefacts, 5 steady images of at least 20 seconds each will be obtained and stored under a random number. Offline blind analysis of each video will be done by two investigators. A previously validated semiquantitative score will be used . It distinguishes between no flow (0), intermittent flow (1), sluggish flow (2), and continuous flow (3). A value is assigned to each individual vessel. The overall score, called the microvascular flow index (MFI), is the average of the individual values. For each patient, the values from 5 videos will be averaged. In addition, vascular density will be quantified as the number of vessels per millimeters squared. To determine heterogeneity of perfusion, the flow heterogeneity index will be calculated as the highest MFI minus the lowest MFI divided by the mean MFI. Finally, the percent of perfused vessels and the total and capillary perfused vascular densities will be calculated. The percent of perfused vessels will be calculated as the number of vessels with flows 2 and 3 divided by the total number of vessels and multiplied by 100. The perfused vascular density will be calculated as the number of vessels multiplied by the fraction of perfused vessels. These quantifications of flow were made per group of vessel diameter: small (capillaries), 10 to 20 μm; medium, 21 to 50 μm; and large, 51 to 100 μm Sample size (number of participants included) 68 patients (34 in each group) Power analysis was performed using Student's t-test for independent samples with MFI as the primary outcome. A previous study demonstrated that MFI during cardiopulmonary bypass was approximately 2.6 + 1. Sample size was calculated to detect a 25% difference in MFI between the two groups with a power of 0.8 and an alpha error of 0.5. A minimum of 62 patients (31 in each group) would be necessary, and this was increased to 68 (34 in each group) to compensate for dropouts.

Statistical analysis Data will expressed as mean + SD, median (range), or frequency as appropriate. Categorical variables will be compared using Chi-square or Fisher's exact test as appropriate. Normally distributed data will be compared using Student's t-test while non-normally distributed data will be compared using Mann-Whitney test or the Kruskal-Wallis test as appropriate. Intergroup comparisons will be done using analysis of variance with repeated measures and post-hoc Dunnett test. A P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged (>18), males and females, undergoing elective coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass (CPB).

Exclusion Criteria:

* Patient refusal.
* Emergency surgeries
* Redo surgeries
* Pregnancy
* Vasculitis
* Inflammation or infection at the study site
* History of allergic reaction to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Microvascular flow index | Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass
  Microcirculation will be studied with side-stream dark field (SDF) imaging (Microscan; MicroVision Medical, Amsterdam, Netherlands) 5 steady images of at least 20 seconds each will be obtained and stored under a random number. Offline blind analysis of each video will be done by two investigators. A previously validated semiquantitative score will be used (15). It distinguishes between no flow (0), intermittent flow (1), sluggish flow (2), and continuous flow (3). A value is assigned to each individual vessel. The overall score, called the microvascular flow index (MFI), is the average of the individual values.

SECONDARY OUTCOMES:
Change in Total vascular density | Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass
  the number of vessels per millimeters squared
Change in perfused vessel density | Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass
  the number of vessels multiplied by the fraction of perfused vessels
Change in proportion of perfused vessel | Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass
  the number of vessels with flows 2 and 3 divided by the total number of vessels and multiplied by 100
Change in Serum lactate | Immediately before starting CBP (T0) , 30 min after initiation of bypass (T1), and 30 min after weaning from bypass
Hemodynamic parameters | Every hour for six hours after induction
  Mean arterial pressure (MAP)
Vasopressor dose | Every hour for six hours after induction

CONTACTS AND LOCATIONS:
Overall Officials: Hisham H Abdel Wahab, MD, Study Chair — Cairo University; Hossam S El-Ashmawi, MD, Principal Investigator — Cairo University; Pierre Z Tawadros, MD, Study Chair — Cairo University; Hassan M Hassan, M.D,FCAI, Study Director — Cairo University
Locations (1):
- Kasr Al-Ainy hospitals , Faculty of medicine , Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koning NJ, Vonk AB, Meesters MI, Oomens T, Verkaik M, Jansen EK, Baufreton C, Boer C. Microcirculatory perfusion is preserved during off-pump but not on-pump cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):336-41. doi: 10.1053/j.jvca.2013.05.026. Epub 2013 Oct 23. PMID 24161555
- [Background] Vellinga NA, Ince C, Boerma EC. Microvascular dysfunction in the surgical patient. Curr Opin Crit Care. 2010 Aug;16(4):377-83. doi: 10.1097/mcc.0b013e32833a0633. PMID 20665963
- [Background] den Uil CA, Lagrand WK, van der Ent M, Jewbali LS, Cheng JM, Spronk PE, Simoons ML. Impaired microcirculation predicts poor outcome of patients with acute myocardial infarction complicated by cardiogenic shock. Eur Heart J. 2010 Dec;31(24):3032-9. doi: 10.1093/eurheartj/ehq324. Epub 2010 Sep 9. PMID 20829210
- [Background] De Backer D, Dubois MJ, Schmartz D, Koch M, Ducart A, Barvais L, Vincent JL. Microcirculatory alterations in cardiac surgery: effects of cardiopulmonary bypass and anesthesia. Ann Thorac Surg. 2009 Nov;88(5):1396-403. doi: 10.1016/j.athoracsur.2009.07.002. PMID 19853081
- [Background] Bauer A, Kofler S, Thiel M, Eifert S, Christ F. Monitoring of the sublingual microcirculation in cardiac surgery using orthogonal polarization spectral imaging: preliminary results. Anesthesiology. 2007 Dec;107(6):939-45. doi: 10.1097/01.anes.0000291442.69337.c9. PMID 18043062
- [Background] Koning NJ, Atasever B, Vonk AB, Boer C. Changes in microcirculatory perfusion and oxygenation during cardiac surgery with or without cardiopulmonary bypass. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1331-40. doi: 10.1053/j.jvca.2013.04.009. Epub 2013 Sep 12. No abstract available. PMID 24035060
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Atasever B, Boer C, Goedhart P, Biervliet J, Seyffert J, Speekenbrink R, Schwarte L, de Mol B, Ince C. Distinct alterations in sublingual microcirculatory blood flow and hemoglobin oxygenation in on-pump and off-pump coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):784-90. doi: 10.1053/j.jvca.2010.09.002. Epub 2010 Nov 5. PMID 21115363
- [Background] Koning NJ, Vonk AB, van Barneveld LJ, Beishuizen A, Atasever B, van den Brom CE, Boer C. Pulsatile flow during cardiopulmonary bypass preserves postoperative microcirculatory perfusion irrespective of systemic hemodynamics. J Appl Physiol (1985). 2012 May;112(10):1727-34. doi: 10.1152/japplphysiol.01191.2011. Epub 2012 Mar 8. PMID 22403352
- [Background] Yuruk K, Almac E, Bezemer R, Goedhart P, de Mol B, Ince C. Blood transfusions recruit the microcirculation during cardiac surgery. Transfusion. 2011 May;51(5):961-7. doi: 10.1111/j.1537-2995.2010.02971.x. Epub 2010 Dec 6. PMID 21133930
- [Background] Savola JM, Virtanen R. Central alpha 2-adrenoceptors are highly stereoselective for dexmedetomidine, the dextro enantiomer of medetomidine. Eur J Pharmacol. 1991 Mar 26;195(2):193-9. doi: 10.1016/0014-2999(91)90535-x. PMID 1678707
- [Background] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Background] Miranda ML, Balarini MM, Bouskela E. Dexmedetomidine attenuates the microcirculatory derangements evoked by experimental sepsis. Anesthesiology. 2015 Mar;122(3):619-30. doi: 10.1097/ALN.0000000000000491. PMID 25313879
- [Background] Yeh YC, Sun WZ, Ko WJ, Chan WS, Fan SZ, Tsai JC, Lin TY. Dexmedetomidine prevents alterations of intestinal microcirculation that are induced by surgical stress and pain in a novel rat model. Anesth Analg. 2012 Jul;115(1):46-53. doi: 10.1213/ANE.0b013e318253631c. Epub 2012 Apr 13. PMID 22504209
- [Background] Boerma EC, Mathura KR, van der Voort PH, Spronk PE, Ince C. Quantifying bedside-derived imaging of microcirculatory abnormalities in septic patients: a prospective validation study. Crit Care. 2005;9(6):R601-6. doi: 10.1186/cc3809. Epub 2005 Sep 22. PMID 16280059
- [Background] den Uil CA, Lagrand WK, Spronk PE, van Domburg RT, Hofland J, Luthen C, Brugts JJ, van der Ent M, Simoons ML. Impaired sublingual microvascular perfusion during surgery with cardiopulmonary bypass: a pilot study. J Thorac Cardiovasc Surg. 2008 Jul;136(1):129-34. doi: 10.1016/j.jtcvs.2007.10.046. Epub 2008 May 2. PMID 18603065